CLINICAL TRIAL: NCT04433546
Title: A Randomized, Double-Blind, Parallel Group Study to Assess the Efficacy and Safety of Once Weekly Subcutaneous Injections of Pemziviptadil (PB1046), a Sustained-Release VIP (Vasoactive Intestinal Peptide) ANalogue, in Hospitalized COVID-19 Patients at HiGh Risk for Rapid Clinical Deterioration and ARDS (PB1046 VANGARD Study)
Brief Title: Pemziviptadil (PB1046), a Long-acting, Sustained Release Human VIP Analogue, Intended to Provide Clinical Improvement to Hospitalized COVID-19 Patients at High Risk for Rapid Clinical Deterioration and Acute Respiratory Distress Syndrome (ARDS).
Acronym: VANGARD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company no longer pursing indication
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0007
Record Dates: First submitted 2020-05-28; First posted 2020-06-16 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Acute Respiratory Distress Syndrome; Coronavirus; Hypoxic Respiratory Failure; Hypoxemic Respiratory Failure; Respiratory Complication; Respiratory Insufficiency; Cardiac Dysfunction; Pneumonia; Pulmonary Edema; Pulmonary Inflammation; Respiratory Failure; Cytokine Storm; COVID 19; SARS-CoV-2; Cardiac Event; Cardiac Complication; Cardiac Failure; Cardiac Infarct
Keywords: Acute Respiratory Distress Syndrome (ARDS); Respiratory distress/failure; COVID
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; Respiratory Insufficiency; Pneumonia; Pulmonary Edema; Cytokine Release Syndrome; COVID-19; Cardiovascular Diseases; Heart Failure; Myocardial Infarction; Dyspnea | interventions — VIP-ELP fusion molecule PB1046

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose (100 mg) Group (Experimental): High: Pemziviptadil (PB1046) 100 mg subcutaneous (SC) weekly for 4 weeks or until hospital discharge
  Interventions: Drug: Pemziviptadil (PB1046)
- Middle Dose (40 mg) Group (Experimental): Middle: Pemziviptadil (PB1046) 40 mg SC weekly for 4 weeks or until hospital discharge
  Interventions: Drug: Pemziviptadil (PB1046)
- Low Dose (10 mg) Control Group (Placebo Comparator): Low Control: Pemziviptadil (PB1046) 10 mg SC weekly for 4 weeks or until hospital discharge
  Interventions: Drug: Low Dose (10 mg) Control

INTERVENTIONS:
Drug: Pemziviptadil (PB1046) — Pemziviptadil (PB1046), Once Weekly Subcutaneous Injection
  Arms: High Dose (100 mg) Group; Middle Dose (40 mg) Group
Drug: Low Dose (10 mg) Control — Pemziviptadil (PB1046), Once Weekly Subcutaneous Injection (10 mg diluted in sodium chloride to match active drug volume)
  Arms: Low Dose (10 mg) Control Group

SUMMARY:
This is a multicenter, randomized, double-blind, parallel group study to investigate the efficacy of pemziviptadil (PB1046) by improving the clinical outcomes in hospitalized COVID-19 patients at high risk for rapid clinical deterioration, acute respiratory distress syndrome (ARDS) and death.

The study will enroll approximately 210 hospitalized COVID-19 patients who require urgent decision-making and treatment at approximately 20 centers in the United States.

DETAILED DESCRIPTION:
The study will consist of a Screening/Pre-treatment period, on-site randomization to study treatment. On Day 0 (Visit 2) subjects who meet inclusion criteria and none of exclusion criteria will receive a weekly subcutaneous injection that will continue once weekly until hospital discharge or for a maximum of 4 weeks during hospitalization, whichever is shorter.

All subjects will be randomized to either a low control (10 mg), middle (40 mg), or high (100 mg) dose of active treatment. If subject is not discharged, they will continue to Day 7, 14, 21 treatments. Pemziviptadil (PB1046) is expected to improve the clinical outcomes of hospitalized COVID-19 subjects with an earlier hospital discharge and improvement in survival.

The duration of hospitalization for each subject will be determined by clinical status independent of study procedures. The estimated duration of the study for each subject, including screening, is approximately 35+7 days. The subjects may be involved up to 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Written or witnessed verbal informed consent from patient or remote legal authorized representative (LAR) or remote family member as permitted by governing local or central Institutional Review Board (IRB)/independent Ethic Committee (IEC).
2. Male or female 18-85 years old hospitalized COVID-19 patients (positive local SARS-CoV2 test)
3. Receiving oxygen (O2) by face mask or nasal cannula/prongs and/or with elevated markers of cardiac injury or dysfunction (hsTnI or NT-proBNP) as assessed by local testing

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Patients considered unsalvageable or expected to expire within 24 hours
2. On mechanical ventilation or imminent need for mechanical ventilation expected in the next 24 hours
3. Evidence of acute end-organ injury in 2 or more organ systems (not including cardiac or pulmonary), such as, renal, hepatic, or CNS injury
4. Receiving another investigational therapy for treatment or prevention of COVID-19-related hypoxemic respiratory failure or ARDS other than antiviral therapy
5. Systolic blood pressure (SBP) < 95 mmHg and/or diastolic blood pressure (DBP) < 50 mmHg or overt symptomatic hypotension during screening
6. Resting heart rate > 110 BPM (beats per minute) during screening
7. Severe chronic renal failure as measured by the estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73m2 using the local laboratory calculation of eGFR.
8. Significant liver dysfunction as measured by any one of the following at screening:

   * ALT (Alanine transaminase) > 3.0 times ULN (upper limit of normal)
   * AST (Aspartate transaminase) > 3.0 times ULN
   * Serum bilirubin ≥ 1.6 mg/dL
9. Any in-patient surgical procedure or hospitalization (defined as > 23 hours) within 30 days of subject screening except for prior hospitalization for COVID-19
10. Known hypersensitivity to study drug or any of the excipients of the drug formulation
11. Pregnant or lactating female subjects
12. Any other condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining informed consent or confound the objectives of study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Time to clinical recovery from initiation of pemziviptadil (PB1046) | 28 days

SECONDARY OUTCOMES:
Time to clinical recovery (being well enough for hospital discharge or returning to normal baseline activity level prior to discharge) | 28 days
Time to hospital discharge | Any time point between injection initiation and Day 28
All-cause mortality | 28 days
Reduction in hospital resource utilization defined as a composite of: total days: in hospital, in ICU, on ventilator, on ECMO, with invasive hemodynamic monitoring, with mechanical circulatory support, and with inotropic or vasopressor therapy | 28 days
  Composite of: Total hospital days, Total ICU days, Total days of ventilator use, Total days of ECMO, Total days of invasive hemodynamic monitoring, Total days of mechanical circulatory support, Total days of inotropic or vasopressor therapy
Time to clinical improvement as defined by reduction of at least 2 points on an 8-category ordinal scale of clinical improvement or discharge from hospital, whichever comes first. | Any time point between injection initiation and Day 28
Change from baseline in cardiac marker troponin I (TrI) | Any time point between injection initiation and Day 35+7
Change from baseline in cardiac marker NT-proBNP/BNP | Any time point between injection initiation and Day 35+7
Change from baseline in TNF alpha | Any time point between injection initiation and Day 35+7
Change from baseline in IL-1 | Any time point between injection initiation and Day 35+7
Change from baseline in IL-6 | Any time point between injection initiation and Day 35+7
Incidence and severity of any treatment emergent adverse events (TEAEs) or serious adverse events (SAEs) as determined by clinical adverse events (AEs) and their relationship to pemziviptadil (PB1046). | Any time point between injection initiation and Day 35+7
Incidence and severity of any treatment emergent adverse events (TEAEs) or serious adverse events (SAEs) as determined by vital signs and their relationship to pemziviptadil (PB1046) | Any time point between injection initiation and Day 35+7
Incidence and severity of any treatment emergent adverse events (TEAEs) or serious adverse events (SAEs) as determined by laboratory results and their relationship to pemziviptadil (PB1046) | Any time point between injection initiation and Day 35+7
Incidence and severity of any treatment emergent adverse events (TEAEs) or serious adverse events (SAEs) as determined by electrocardiogram (ECG) abnormalities and their relationship to pemziviptadil (PB1046) | Any time point between injection initiation and Day 35+7
Incidence and severity of any treatment emergent adverse events (TEAEs) or serious adverse events (SAEs) as determined by incidence of anti-drug antibodies and their relationship to pemziviptadil (PB1046) | Any time point between injection initiation and Day 35+7

OTHER OUTCOMES:
Impact on invasive hemodynamic parameters as measured by pulmonary artery pressure if patients require right-heart catherization | Any time point between injection initiation and Day 35+7
Impact on invasive hemodynamic parameters as measured by cardiac output if patients require right-heart catherization | Any time point between injection initiation and Day 35+7
Incidence of multi-system organ failure (MSOF) | Any time point between injection initiation and Day 35+7
Number of multi-system organ failure (MSOF) free days | Any time point between injection initiation and Day 35+7
Number of subjects requiring extracorporeal membrane oxygenation (ECMO) | Any time point between injection initiation and Day 35+7
Change in circulating ferritin | Any time point between injection initiation and Day 35+7
Change in circulating D-dimer | Any time point between injection initiation and Day 35+7
Change in liver function | Any time point between injection initiation and Day 35+7
Change in other blood chemistry | Any time point between injection initiation and Day 35+7
Change in hematology | Any time point between injection initiation and Day 35+7
Change in inflammatory markers | Any time point between injection initiation and Day 35+7
Change in coagulation markers | Any time point between injection initiation and Day 35+7
Percent of clinical failure | Any time point between injection initiation and Day 35+7

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Baptist Health Research Institute, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Adventist Healthcare White Oak Medical Center, Silver Spring, Maryland